CLINICAL TRIAL: NCT03192449
Title: Serum Pharmacokinetic Disposition and Urinary Excretion of Albendazole and Its Metabolites in Non-infected Human Volunteers.
Brief Title: Serum Pharmacokinetic Disposition and Urinary Excretion of Albendazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Nacional de Salta (Other)
Collaborators: CIVETAN CONICET, Facultad de Ciencias Veterinarias, UNCPBA. Tandil (Unknown)
Responsible Party: Principal Investigator, Alejandro Krolewiecki, Principal Investigator, Universidad Nacional de Salta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIVETAN-IIET-ALB01
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Soil Transmitted Helminthiasis; Neglected Tropical Diseases
MeSH Terms: conditions — Neglected Diseases | interventions — Albendazole

STUDY DESIGN:
Intervention Model Description: Pharmacokinetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albendazole 400mg p.o. single dose (Experimental): Volunteers receive 1 tablet albendazole 400mg (GSK) fasting.
  Interventions: Drug: Albendazole.

INTERVENTIONS:
Drug: Albendazole. — Single dose 400mg orally

SUMMARY:
Mass drug administration (MDA) of albendazole (ABZ) to school-age and pre-school-age children is the currently recommended strategy for controlling soil-transmitted helminthiasis (STH) in endemic areas. Recent mathematical modelling suggests that community-wide MDA will be required in order to interrupt transmission of STH. DEWORM3 aims to determine the feasibility of eliminating STH through expanded and intensified MDA strategies. In order to ensure rigorous trial results, it is crucial that the definition of such MDA coverage is informed by unbiased, empirical data. The Centro de Investigación Veterinaria de Tandil (CIVETAN) and Instituto de Investigaciones en Enfermedades Tropicales Universidad Nacional de Salta collaborate on scientific research related to pharmacokinetic studies of ABZ.

This proposal describes the request for funding from DEWORM3 to conduct a study of the serum pharmacokinetic characteristics and urinary excretion of ABZ and its metabolites in non-infected human volunteers to better understand the use of urinary analysis of ABZ as a measure of MDA adherence in the context of DEWORM3.

DETAILED DESCRIPTION:
Objective 1.To characterize the plasma disposition kinetics of ABZ and its main metabolites (ABZ sulphoxide and ABZ sulphone) in non-infected human volunteers.

Objective 2. To characterize the pattern of albendazole (ABZ) and its main metabolites (ABZ sulphoxide and ABZ sulphone) urinary excretion in non-infected human volunteers.

Objective 3. To determine the optimal and the longest period time after treatment where either ABZ and/or its metabolites can be measured in urine as an indirect assessment of an individual's adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Weight between 45 and 75 Kg.
2. Physical exam without significant abnormal findings.

Exclusion Criteria:

1. Intake of ABZ or other benzimidazole drugs within the last 30 days.
2. Malabsorption or other GI syndromes that could compromise the tolerability or absorption of ABZ.
3. History of hypersensitivity or intolerance to ABZ or its inactive ingredients.
4. Acute clinical conditions.
5. Pregnancy or breast feeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Albendazole in urine | Up to 72 hours
  Urinary excretion of albendazole (ABZ) and its main metabolites (ABZ sulphoxide and ABZ sulphone) in non-infected human volunteers. PK parameters (Cmax, AUC, Tmax) from levels measured through HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro J Krolewiecki, MD/PhD, Study Director — Universidad Nacional de Salta

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer review journal

REFERENCES:
- [Derived] Ceballos L, Krolewiecki A, Juarez M, Moreno L, Schaer F, Alvarez LI, Cimino R, Walson J, Lanusse CE. Assessment of serum pharmacokinetics and urinary excretion of albendazole and its metabolites in human volunteers. PLoS Negl Trop Dis. 2018 Jan 18;12(1):e0005945. doi: 10.1371/journal.pntd.0005945. eCollection 2018 Jan. PMID 29346367